CLINICAL TRIAL: NCT04612816
Title: Live Stream of Emergency Ultrasound to Improve Diagnostics in Prehospital Medical Care: a Feasibility Study
Brief Title: Live Stream of Ultrasound in Prehospital Medical Care
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Martina Loinger, Researcher, Medical University of Vienna
Other Study IDs: Prehospital Ultrasound LBI/MUV
Record Dates: First submitted 2020-10-20; First posted 2020-11-03 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Ultrasound
Keywords: echocardiography; emergency medicine; telemedicine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Prehospital ultrasound — Feasibility of real time PEU transmission in a university affiliated preclinical emergency system.

SUMMARY:
Prehospital emergency ultrasound (PEU) is being increasingly used in different preclinical emergency systems across the world. Ultrasound examinations in emergency situations, however, remain challenging even in the hospital setting despite the availability of standardized approaches such as Focused Assessment with Sonography for Trauma (FAST). Preclinical circumstances further complicate the adequate execution of an additional diagnostic tool such as PEU on the scene or inside a medical emergency vehicle. Furthermore, rapid translation of ultrasound findings into meaningful therapeutic consequences is considerably demanding in an environment of limited resources. If focused PEU is correctly used and patients' condition allows emergency doctors a careful ultrasound examination, it is possible to differentiate life-threatening diagnoses. PEU should be implemented in the management of emergency patients affected by trauma, cardiac arrest/shock or respiratory problems. To date it is unclear whether PEU results in improved outcome.

Some emergency cases present difficult challenges in the prehospital ultrasound examination. Portable devices designed for PEU suggest the possibility of increasing the use of ultrasound "in the field". However, to the investigator's knowledge, opportunities for real-time consultation with a second specialist including live transmission of the ultrasound picture are not being provided at any preclinical emergency facility.

DETAILED DESCRIPTION:
Aim 1:

Feasibility of real time prehospital emergency ultrasound (PEU) transmission in a university affiliated preclinical emergency system.

Aim 2:

Identify obstacles for PEU transmission including a real time consultation of an ultrasound expert.

Hypothesis:

We expect that live streaming of emergency ultrasound images in order to allow a second opinion could improve diagnostics of life threatening conditions and help us to improve patients' safety by digital health. The use of PEU is feasible and safe.

ELIGIBILITY:
Inclusion Criteria:

Emergency patients affected by:

* trauma
* cardiac arrest/shock
* respiratory problems

Exclusion Criteria:

* Patients rejection.
* Legal representative's rejection.

Ages: 18 Years to 116 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PEU should be implemented in the management of emergency patients affected by trauma, cardiac arrest/shock or respiratory problems.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Quality of PEU live stream. | 3 Months
  Numerical scale (1-10; 1 = best, 10 = poor)

SECONDARY OUTCOMES:
Identify obstacles for PEU transmission including a real time consultation of an ultrasound expert. | 3 Months
  Expert available on time? Communication? Duration of ultrasound examination? Duration of live stream? Delay by PEU transmission? Emergency duration with/without PEU transmission Technical problems?
Identify obstacles for PEU transmission including a real time consultation of an ultrasound expert. | 3 Months
  Communication?
Identify obstacles for PEU transmission including a real time consultation of an ultrasound expert. | 3 Months
  Duration of ultrasound examination?
Identify obstacles for PEU transmission including a real time consultation of an ultrasound expert. | 3 Months
  Duration of live stream?
Identify obstacles for PEU transmission including a real time consultation of an ultrasound expert. | 3 Months
  Delay by PEU transmission?
Identify obstacles for PEU transmission including a real time consultation of an ultrasound expert. | 3 Months
  Emergency duration with/without PEU transmission technical problems?

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna - Division of General Anaesthesia and Intensive Care Medicine, Vienna, Austria

REFERENCES:
- [Background] Botker MT, Jacobsen L, Rudolph SS, Knudsen L. The role of point of care ultrasound in prehospital critical care: a systematic review. Scand J Trauma Resusc Emerg Med. 2018 Jun 26;26(1):51. doi: 10.1186/s13049-018-0518-x. PMID 29940990
- [Background] van der Weide L, Popal Z, Terra M, Schwarte LA, Ket JCF, Kooij FO, Exadaktylos AK, Zuidema WP, Giannakopoulos GF. Prehospital ultrasound in the management of trauma patients: Systematic review of the literature. Injury. 2019 Dec;50(12):2167-2175. doi: 10.1016/j.injury.2019.09.034. Epub 2019 Sep 28. PMID 31627899
- [Background] Scharonow M, Weilbach C. Prehospital point-of-care emergency ultrasound: a cohort study. Scand J Trauma Resusc Emerg Med. 2018 Jun 18;26(1):49. doi: 10.1186/s13049-018-0519-9. PMID 29914554
- [Background] Ketelaars R, Reijnders G, van Geffen GJ, Scheffer GJ, Hoogerwerf N. ABCDE of prehospital ultrasonography: a narrative review. Crit Ultrasound J. 2018 Aug 8;10(1):17. doi: 10.1186/s13089-018-0099-y. PMID 30088160
- [Background] Marsh-Feiley G, Eadie L, Wilson P. Telesonography in emergency medicine: A systematic review. PLoS One. 2018 May 3;13(5):e0194840. doi: 10.1371/journal.pone.0194840. eCollection 2018. PMID 29723198
- [Background] Schmid M, Dodt C. [Emergency lung ultrasound]. Med Klin Intensivmed Notfmed. 2018 Nov;113(8):616-624. doi: 10.1007/s00063-018-0485-z. Epub 2018 Oct 10. German. PMID 30306189
- [Derived] Hermann M, Hafner C, Scharner V, Hribersek M, Maleczek M, Schmid A, Schaden E, Willschke H, Hamp T. Remote real-time supervision of prehospital point-of-care ultrasound: a feasibility study. Scand J Trauma Resusc Emerg Med. 2022 Mar 24;30(1):23. doi: 10.1186/s13049-021-00985-0. PMID 35331304